CLINICAL TRIAL: NCT00186576
Title: Non-Myeloablative Allogeneic Hematopoietic Cell Transplantation for Treatment of Myelodysplastic Syndromes and Myeloproliferative Disorders (Except CML)
Brief Title: Non-Myeloablative Allogeneic Transplant for Myelodysplastic Syndromes and Myeloproliferative Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Ginna Laport, Stanford University School of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMT128; 75826; BMT128; NCT00186576; NCT00052546 (obsolete NCT alias)
Record Dates: First submitted 2005-09-14; First posted 2005-09-16 (Estimated); Last update posted 2010-10-14 (Estimated); Status verified 2010-10

CONDITIONS: Myelodysplastic Syndromes; Myeloproliferative Disorders; Blood and Marrow Transplant (BMT); Myelodysplastic Syndromes (MDS); Myeloproliferative Disorders (MPD)
MeSH Terms: conditions — Myelodysplastic Syndromes; Myeloproliferative Disorders

INTERVENTIONS:
Procedure: nonmyeloablative allogeneic hematopoietic cell transplant

SUMMARY:
To improve survival outcomes for patients with MDS and MPD with a nonmyeloablative allogeneic hematopoietic cell transplant.

DETAILED DESCRIPTION:
Non-Myeloablative Allogeneic Hematopoietic Cell Transplantation for Treatment of Myelodysplastic Syndromes and Myeloproliferative Disorders (Except CML)

ELIGIBILITY:
Inclusion Criteria:- Myelodysplastic Syndromes

* Myeloproliferative Disorders
* HLA matched donor available Exclusion Criteria:- organ dysfunction
* HIV positive

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2001-12; Primary Completion 2004-03 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Efficacy of transplant | 1 year

SECONDARY OUTCOMES:
safety profile of nonmyeloablative transplant, graft versus host disease, graft rejection, non-relapse mortality, use of donor lymphocyte infusion | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ginna Laport, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Result] Laport GG, Sandmaier BM, Storer BE, Scott BL, Stuart MJ, Lange T, Maris MB, Agura ED, Chauncey TR, Wong RM, Forman SJ, Petersen FB, Wade JC, Epner E, Bruno B, Bethge WA, Curtin PT, Maloney DG, Blume KG, Storb RF. Reduced-intensity conditioning followed by allogeneic hematopoietic cell transplantation for adult patients with myelodysplastic syndrome and myeloproliferative disorders. Biol Blood Marrow Transplant. 2008 Feb;14(2):246-55. doi: 10.1016/j.bbmt.2007.11.012. PMID 18215785
- [Derived] Cooper JP, Storer BE, Granot N, Gyurkocza B, Sorror ML, Chauncey TR, Shizuru J, Franke GN, Maris MB, Boyer M, Bruno B, Sahebi F, Langston AA, Hari P, Agura ED, Lykke Petersen S, Maziarz RT, Bethge W, Asch J, Gutman JA, Olesen G, Yeager AM, Hubel K, Hogan WJ, Maloney DG, Mielcarek M, Martin PJ, Flowers MED, Georges GE, Woolfrey AE, Deeg JH, Scott BL, McDonald GB, Storb R, Sandmaier BM. Allogeneic hematopoietic cell transplantation with non-myeloablative conditioning for patients with hematologic malignancies: Improved outcomes over two decades. Haematologica. 2021 Jun 1;106(6):1599-1607. doi: 10.3324/haematol.2020.248187. PMID 32499241